CLINICAL TRIAL: NCT04402749
Title: The Incidence of Perioperative Pulmonary Embolism in Patients With Renal Carcinoma Undergoing Nephrectomy
Brief Title: The Incidence of Pulmonary Embolism During Nephrectomy
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_2
Record Dates: First submitted 2020-05-07; First posted 2020-05-27 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Embolism; Renal Cell Carcinoma; Nephrectomy
MeSH Terms: conditions — Pulmonary Embolism; Carcinoma, Renal Cell | interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nephrectomy: Patients underwent nephrectomy
  Interventions: Other: Nephrectomy

INTERVENTIONS:
Other: Nephrectomy — Patients underwent nephrectomy

SUMMARY:
Patients with renal carcinoma was reported at high incidence of perioperative pulmonary embolism from current study. The investigators aimed to determine the incidence and outcome of this group of patient in the tertiary-care, university hospital and the rate of intraoperative transesophageal echocardiography utility and outcome.

DETAILED DESCRIPTION:
Perioperative pulmonary embolism (PE) is the serious adverse event leading to major morbidity and mortality. The incidence of PE during urologic surgery was previously report at 0.9 - 1.1% with mortality rate less than 2%. But the recent study by Fukazawa et al report the incidence of PE was 11% in renal cancer patients underwent nephrectomy with mortality rate as high as 33%. The risk factors associated with PE included major surgery, cancer, arrhythmia, massive bleeding and level of tumor thrombus in inferior vena cava.

Transesophageal echocardiography (TEE) is a very helpful intraoperative monitoring tool in major, non-cardiac surgery to detect emboli and guide the hemodynamic management in severely unstable patients. But it requires sophisticate machine and well-trained operator, the rate of utilisation was still limited.

The investigators aimed to determine the incidence of perioperative PE in renal cancer patients undergoing nephrectomy. the secondary outcomes include risk factors associated with perioperative PE, clinical outcomes, the rate of TEE utilization in this operation and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with renal cancer undergoing nephrectomy

Exclusion Criteria:

* Patients with incomplete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every adult patients with renal carcinoma underwent nephrectomy will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The incidence of intraoperative PE of renal cancer patient undergoing nephrectomy | intraoperative period
  Pulmonary embolism
  * Clinical suspicious:Systolic blood pressure < 90 mmHg without other reasonable causes, partial pressure of oxygen in artery < 80 mmHg
  * Confirmed diagnosis: intraoperative TEE (direct demonstration of PE or indirect signs of PE), CT angiography, perfusion lung scan

SECONDARY OUTCOMES:
The incidence of postoperative PE of renal cancer patient undergoing nephrectomy | until 7 days after surgery
  Pulmonary embolism
  * Clinical suspicious:Systolic blood pressure < 90 mmHg without other reasonable causes, partial pressure of oxygen in artery < 80 mmHg
  * Confirmed diagnosis: intraoperative TEE (direct demonstration of PE or indirect signs of PE), CT angiography, perfusion lung scan
Length of stay | 7 days after surgery
  * Hospital stay
  * ICU stay
Number of patients with postoperative organ dysfunction | 7 days after surgery
  Organ dysfunction
  * acute kidney injury
  * acute respiratory distress syndrome
Rate of TEE utilization | 7 days after surgery
  TEE utilization
  * for monitoring (use when the case begins)
  * for rescue (use when unexplained hypotension or hemodynamic collapsed)
Mortality rate at 30 days postoperative | 30 days after surgery
  Patients death after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aphichat Suphathamwit, M.D., Principal Investigator — Faculty of Medicine Siriraj Hospital, Mahidol University, THAILAND
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desciak MC, Martin DE. Perioperative pulmonary embolism: diagnosis and anesthetic management. J Clin Anesth. 2011 Mar;23(2):153-65. doi: 10.1016/j.jclinane.2010.06.011. PMID 21377083
- [Result] Cisek LJ, Walsh PC. Thromboembolic complications following radical retropubic prostatectomy. Influence of external sequential pneumatic compression devices. Urology. 1993 Oct;42(4):406-8. doi: 10.1016/0090-4295(93)90369-l. PMID 8212439
- [Result] Pettus JA, Eggener SE, Shabsigh A, Yanke B, Snyder ME, Serio A, Vickers A, Russo P, Donat SM. Perioperative clinical thromboembolic events after radical or partial nephrectomy. Urology. 2006 Nov;68(5):988-92. doi: 10.1016/j.urology.2006.06.026. PMID 17113889
- [Result] Fukazawa K, Fong CT, Gologorsky E. Inferior Vena Cava Tumor Thrombus Dynamics and Perioperative Pulmonary Embolism: A Single-Center Experience. J Cardiothorac Vasc Anesth. 2019 Oct;33(10):2728-2734. doi: 10.1053/j.jvca.2019.03.011. Epub 2019 Mar 15. PMID 31072702